CLINICAL TRIAL: NCT05822856
Title: Gut Microbiota: a Player in the Patients Pain's Sensitization With Rheumatoid Arthritis?
Brief Title: Gut Microbiota: a Player in Chronic Pain in Patients With Rheumatoid Arthritis?
Acronym: MiSenDol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0385
Record Dates: First submitted 2023-04-07; First posted 2023-04-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis; Fibromyalgia
Keywords: Rheumatoid Arthritis; intestinal microbiota; Faecalibacterium; pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Fibromyalgia; Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and intestinal microbiota (stool) samples taken in the framework of the research will constitute a serum library and a bank of intestinal microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with RA without inflammation with persistent chronic pain: Blood sampling, faeces collection, questionnaires, tactile sensitivity, sensorial tests
  Interventions: Other: Blood sampling and others interventions
- Patients with an active RA (in inflammatory flare): Blood sampling, faeces collection, questionnaires, tactile sensitivity, sensorial tests
  Interventions: Other: Blood sampling and others interventions
- Patients with RA in remission without pain: Blood sampling, faeces collection, questionnaires, tactile sensitivity, sensorial tests
  Interventions: Other: Blood sampling and others interventions
- fibromyalgia patients: Blood sampling, faeces collection, questionnaires, tactile sensitivity, sensorial tests
  Interventions: Other: Blood sampling and others interventions
- Control subjects: healthy volunteers: Blood sampling, faeces collection, questionnaires, tactile sensitivity, sensorial tests
  Interventions: Other: Blood sampling and others interventions

INTERVENTIONS:
Other: Blood sampling and others interventions — Blood sampling, faeces collection, questionnaires, tactile sensitivity, sensorial tests

SUMMARY:
Although rheumatoid arthritis (RA) treatments are very effective in reducing inflammation, chronic pain persists in 20 to 30% of patients.

The intestinal microbiota can participate on the pain pathways and a decrease in Faecalibacterium has been associated with chronic pain and chronic fatigue. RA patients have an altered gut microbiota or dysbiosis. Among the bacteria that are most often differentially represented between RA and control, Faecalibacterium, was also found less abundant in RA patients.

The composition of the gut microbiota has never been evaluated in relation to the clinical phenotype of RA patients and in particular to the presence of a diffuse pain. In this study, investigators will test whether the gut microbiota of RA patients, and in particular the decrease of Faecalibacterium, would promote pain sensitization phenomena, and thus, chronic pain despite the control of joint inflammation.

DETAILED DESCRIPTION:
There are currently many treatments available for patients with rheumatoid arthritis (RA). Although these treatments are very effective on inflammation, chronic pain persists in 20 to 30% of patients, even though clinical and biological remission seems to have been achieved, greatly reducing their daily quality of life. They are characterized in particular by a global lowering of pain thresholds, with a clinical picture of secondary fibromyalgia. Indeed, it seems that RA patients present central and peripheral hypersensitization of nociceptors, abnormalities in central pain processing and a defect in top-down inhibitory pain control mechanisms. It is also possible that RA patients with these inflammation-dissociated polyalgic pictures have a different pathophysiology of their disease than those with inflammation-only pain. A growing body of work shows that the gut microbiota (GM) affects pain pathways at multiple levels through the gut-brain axis. This axis relies, among others, on the afferent pathways of the vagus nerve. The microbiota modulates the activity of the vagus nerve by releasing neurotransmitters (gamma-aminobutyric acid, dopamine), by modulating immune cells (cytokines), by modulating the secretions of enteroendocrine cells (serotonin, cholecystokinins, glucagon-like peptide-1, peptide XY) or by releasing metabolites such as short-chain fatty acids, including butyrate. The latter is known to bind to several functional receptors present on vagal afferents. A decrease in Faecalibacterium has been associated with chronic pain and chronic fatigue.

RA is associated with dysbiosis of the gut microbiota, i.e. a change in the composition of the gut flora . Among the bacteria that are most often differentially represented between RA and control, Fecal bacteria are also less abundant in RA patients. The research team has conducted several experiments that clearly confirm the hypothesis that the microbiota of RA patients acts differently on the gut-brain axis than that of healthy subjects. Indeed, it is known that these RA patients present a defect in the control of parasympathetic activity and a link between dysbiosis of the GM and alteration of the autonomous nervous system (ANS) has already been shown in several pathologies. Considering that the GM is altered in RA and that alterations in the GM can modulate the ANS, the research team therefore hypothesized that the GM of RA patients is capable of altering cardiovascular function and particularly autonomic function. To demonstrate the role of the GM in ANS alterations, a mouse model with humanized microbiota by fecal microbiota transplantation (FMT) of RA patients or healthy subjects (age- and sex-matched controls) was developed and the research team showed that transfer of gut microbiota from RA patients toof mice previously treated with antibiotics alters the autonomic control of cardiac rhythm. Indeed, a decrease in vagal activity, objectified by the analysis of heart rate variability was observed, unpublished data. This confirms our hypothesis that the microbiota of RA patients acts differently on the gut-brain axis than that of healthy subjects. There is therefore a strong rationale for thinking that the microbiota of these patients could influence the central sensitization and control of pain and that RA patients with a fibromyalgia profile have a different microbiota from others.

Bacterial extracellular vesicles (EVs) are important vectors of communication between the gut microbiota and its host. They are the subject of increasing attention and could participate in the gut-brain axis. Indeed, some pathogenic EVs participate in the alteration of the intestinal barrier, pass into the bloodstream and can therefore act remotely from the intestine. Moreover, it has been shown that some bacteria (e.g. A. muciniphila and Faecalibacterium Prausnitzii) modulate the intestinal serotonin system mainly via their EVs. However, our preliminary experiments with stool transfer from RA patients suggest that serotonin (5-hydroxytryptamine 5 HT) is altered, as the research team showed that its expression is decreased in the intestine of mice transplanted with stool from RA patients (unpublished).

Hypothesis: RA patients have an altered gut microbiota or dysbiosis. Among the bacteria that are most often differentially found between RA and control, Faecalibacterium are less abundant in RA patients and a decrease in Faecalibacterium has also been associated with chronic pain patterns . The research team therefore hypothesizes that the intestinal microbiota of RA patients, and in particular the decrease in Faecalibacterium, would promote pain sensitization phenomena, the lack of top-down inhibitory control, and thus chronic pain despite the control of joint inflammation.

To test this hypothesis, the investigating team will compare the composition of the gut microbiota of patients with RA in inflammatory flare, RA in pain-free remission, RA without inflammation with chronic pain, healthy subjects without pain, and patients with fibromyalgia without inflammatory rheumatism. Microbial analysis by 16S ribosomal RNA gene sequencing and quantification of major microbiota-derived fecal metabolites (including short-chain fatty acids and tryptophan derivatives and vesicles

Next, investigators will also functionally evaluate the impact of the gut microbiota on pain sensitization. For this purpose, the research team will use in vitro experimental models (intestinal barrier models (Caco2) and neurons of vagal afferents (primary cultures obtained from murine jugular and nuchal ganglia). In an in vivo study, some faeces samples will be used to humanize the mouse microbiota and then evaluate the impact on tactile sensitivity (Von-Frey).

ELIGIBILITY:
Inclusion Criteria:

For all :

- Age ≥ 18 years old

For A1 Group (3 groups of RA patients of 25 patients each):

- Subject with Rheumatoid Arthritis (RA) meeting the American College of Rheumatology / European League Against Rheumatism ACR/EULAR 2010 criteria, without disease-modifying treatment or with conventional treatment initiated for at least 3 months (at stable dosage for more than 6 weeks)

For A1-1 group : active RA

* DAS28>3.2 with increased CRP (> laboratory standard),
* VAS (Visual Analogic Scale)>5/10 with no other explanation than inflammatory rheumatism

For A1-2 group : RA without inflammation with persistent chronic pain (>3 months) despite control of inflammation and no other identified cause:

* no swollen joint,
* CRP normal (< laboratory standard),
* VAS>5/10

For A1-3 groupe : RA in remission without pain:

* DAS28 ≤2.6,
* no swollen joint,
* CRP normal (< laboratory standard),
* VAS≤2/10

For A2 Group (1 group of 25 Fibromyalgia patients):

* Subjects with Fibromyalgia meeting 2016 diagnostic criteria
* VAS>5/10
* FIRST (FIbromyalgia Rapid Screening Tool) ≥5

For A3 Group (1 group of 25 healthy subjects ):

* healthy and pain-free controls subjects with no progressive disease,
* VAS≤2/10,
* FIRST =0

Exclusion Criteria:

* biological therapy for RA: within the previous year for rituximab, within < 4 intervals between anti-TNF, anti-IL6R, or CTLA4-Ig injections and within the previous 15 days for JAKi (JAK inhibitor)
* Corticosteroids > 10 mg/d per os at inclusion
* Corticosteroids > 20 mg/d per os or bolus within 15 days prior to inclusion
* Non-steroidal anti-inflammatory drugs (NSAIDs) and pain medication in the previous week
* Current oral anti-diabetic or proton pump inhibitor (PPI) therapy
* Antibiotic therapy in the previous 3 months
* Infection, cancer in the last 5 years prior to inclusion
* History of other systemic inflammatory/autoimmune diseases
* Not affiliated to a social security
* Patient unwilling or unable to give consent: patient under guardianship or conservatorship,
* Mentally impaired, dementia, language barrier
* Patient under court protection
* Pregnant or breastfeeding woman
* Refusal of written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population with a painful pathology (RA and fibromyalgia) compared to a non-painful population (RA and healthy subjects)
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of the frequency of intestinal Faecalibacterium between : - inflammation-free RA with persistent chronic pain patients and - RA remission pain-free patients | Baseline
  Comparison of the frequency of intestinal Faecalibacterium assessed by 16S RNA sequencing from patient stool samples collected in OMNIGene-Gut collection tubes

SECONDARY OUTCOMES:
comparison of the frequency of intestinal Faecalibacterium between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Frequency of different families, genera, species, alpha diversity evaluated by Shannon index and bacterial richness
comparison of the frequency of intestinal Faecalibacterium between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Frequency of different families, genera, species, alpha diversity evaluated by Shannon index and bacterial richness
comparison of the frequency of intestinal Faecalibacterium between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Frequency of different families, genera, species, alpha diversity evaluated by Shannon index and bacterial richness
comparison of the metabolites from the microbiota between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Concentrations of short chain fatty acids and tryptophan metabolites evaluated by Nuclear magnetic resonance (NMR) in the feces
comparison of the metabolites from the microbiota between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Concentrations of short chain fatty acids and tryptophan metabolites evaluated by Nuclear magnetic resonance (NMR) in the feces
comparison of the metabolites from the microbiota between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Concentrations of short chain fatty acids and tryptophan metabolites evaluated by Nuclear magnetic resonance (NMR) in the feces
Comparison of markers of intestinal permeability between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Quantification of intestinal permeability markers (ZO-1, LBP, CD14-soluble, iFABP) in the serum of the participants by ELISA technique
Comparison of markers of intestinal permeability between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Quantification of intestinal permeability markers (ZO-1, LBP, CD14-soluble, iFABP) in the serum of the participants by ELISA technique
Comparison of markers of intestinal permeability between: - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Quantification of intestinal permeability markers (ZO-1, LBP, CD14-soluble, iFABP) in the serum of the participants by ELISA technique
comparison of markers inflammation (CRP, pro-inflammatory cytokines) between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Quantification of inflammation marker (CRP, pro-inflammatory cytokines) in the serum.
comparison of markers inflammation (CRP, pro-inflammatory cytokines) between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Quantification of inflammation marker (CRP, pro-inflammatory cytokines) in the serum.
comparison of markers inflammation (CRP, pro-inflammatory cytokines) between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Quantification of inflammation marker (CRP, pro-inflammatory cytokines) in the serum.
Comparison of the neurotrophic marker BDNF between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Quantification of the neurotrophic marker BDNF in the blood.
Comparison of the neurotrophic marker BDNF between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Quantification of the neurotrophic marker BDNF in the blood.
Comparison of the neurotrophic marker BDNF between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Quantification of the neurotrophic marker BDNF in the blood.
comparison of fecal calprotectin between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Quantification of fecal calprotectin.
comparison of fecal calprotectin between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Quantification of fecal calprotectin.
comparison of fecal calprotectin between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Quantification of fecal calprotectin.
comparison of the tactile sensitivity and the Visual Analogue Scale (VAS) pains between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves)
comparison of the tactile sensitivity and the Visual Analogue Scale (VAS) pains between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves)
comparison of the tactile sensitivity and the Visual Analogue Scale (VAS) pains between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves)
To investigate the association between tactile sensitivity by the Von-Frey filament technique, bacteria, bacterial metabolites and biomarkers | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves) study of the bacterial population by 16s RNA sequencing determination of bacterial metabolites by Magnetic resonance neurography (MRN) determination of blood biomarkers (intestinal permeability, inflammation and BDNF)
comparison of the central pain sensitivity (QST) data between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - active RA patients | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves)
comparison of the central pain sensitivity (QST) data between : - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - healthy subjects | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves)
comparison of the central pain sensitivity (QST) data between: - RA in remission without pain patients and RA without inflammation with persistant chronic pain patients - patients with fibromyalgia | Baseline
  Tactile sensitivity using the Von-frey filament technique in front of the affected joints in RA (metacarpophalangeal) and at a distance from the joints (forearms and calves)
comparison of the Extracellular Vesicles from microbiota (fecal and circulating). | Baseline
  Isolation, Quantification and Characterization of extracellular vesicles resulting from the interaction host / microbiota interaction
Functional evaluation in an experimental models of the effect of the intestinal microbiota on pain sensitization | Baseline
  impact on in vitro study models of the intestinal barrier (Caco2) and on vagal afferents neurons (primary cultures))
  impact on in vitro intestinal barrier study models (Caco2) and on vagal afferent neurons (primary cultures obtained from murine jugular and nodes) exposed to supernatants from the stools of different patients and to metabolites identified in the comparison of patients' stools. We will also expose them to circulating extracellular vesicles (EVs) in the circulation and in the stool
In vivo (mice) verification of the effect of microbiota on pain. | Baseline
  Transfer of stool samples from patients in a mouse model then a comparison of tactile sensitivity by the Von-frey filament technique

CONTACTS AND LOCATIONS:
Overall Officials: Claire I DAIEN, MD-PhD, Study Director — Centre Hospitalier Universitaire de Montpellier Montpellier
Locations (1):
- CHU montpellier - department of rheumatology, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided